CLINICAL TRIAL: NCT06395285
Title: A Phase Ib, Open-Label Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Orally Administered DF-003 in ROSAH Syndrome Patients
Brief Title: Evaluating the Safety and Tolerability of Orally Administered DF-003 in ROSAH Syndrome Patients
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Yao Yuan Biotechnology Ltd. (also known as Drug Farm) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DF-003-1002
Record Dates: First submitted 2024-04-25; First posted 2024-05-02 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: ROSAH
Keywords: ROSAH syndrome; alpha-protein kinase 1; cone-rod dystrophy; macular edema; papillary edema; retinal dystrophy; uveitis; T237M
MeSH Terms: conditions — Cone-Rod Dystrophies; Macular Edema; Retinal Dystrophies; Uveitis

STUDY DESIGN:
Intervention Model Description: ROSAH syndrome patients will receive oral (PO) doses of DF-003 once daily (QD) for a duration of 28 days (4 weeks). In this study, 8 patients will be evaluated in one cohort. The cohort will have a minimum of 6 patients. Additional patients (maximum of 12 patients) may be enrolled in the event of insufficient data.
  Patients will receive loading doses of 140 mg on Days 1, 2, and 3, followed by a maintenance dose of 45 mg QD starting on Day 4 through Day 28. Individual dose modification is not allowed in this study. If the overall cohort dose needs modification, this will be determined based on review of all available safety and pharmacokinetics (PK) data from this study.
Masking Description: As this is an open label study, there are no blinding requirements for safety data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- DF-003 (Experimental): Oral (PO) doses of 140 mg DF-003 on Days 1, 2, and 3 followed by a maintenance dose of 45 mg DF-003 once daily (QD) starting on Day 4 through Day 28. DF-003 will be administered PO with approximately 240 mL of water in the morning once daily for 28 consecutive days.
  Interventions: Drug: DF-003

INTERVENTIONS:
Drug: DF-003 — 140 mg on Days 1, 2, and 3 followed by a maintenance dose of 45 mg QD starting on Day 4 through Day 28. DF-003 will be administered PO with approximately 240 mL of water in the morning once daily for 28 consecutive days.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of DF-003 in retinal dystrophy, optic nerve edema, splenomegaly, anhidrosis, and migraine headache (ROSAH) syndrome patients.

DETAILED DESCRIPTION:
This is a Phase Ib open-label, single-arm, single-dose study that will be conducted in up to 12 ROSAH syndrome patients. The study will investigate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of DF-003 (study drug). DF-003 will be administered orally (PO), once daily (QD) for 28 days (4 weeks). Patients will be followed up for 8 weeks after administration of the last dose of study drug.

A total of 8 patients will be evaluated in one cohort. The cohort will have a minimum of 6 patients. Additional patients (maximum of 12 patients) may be enrolled in the event of insufficient data after a review of safety data by the Study Safety Committee. Patients will receive loading doses of 140 mg DF-003 on Days 1, 2, and 3, followed by a maintenance dose of 45 mg DF-003 starting on Day 4 through Day 28. Individual dose modification is not allowed in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Sufficient understanding of the purpose and procedures required for the study.
2. Body mass index (BMI) of 18.0 to 35.0 kg/m2, inclusive.
3. Genetic testing for ALPK1 mutations that has been shown to be associated with ROSAH syndrome (e.g. T237M or Y254C, or T237A mutations).
4. Signs of uveitis (anterior and/or posterior) in the eye (e.g. macula edema, optic nerve edema, retinal vasculitis, or retinal vascular leakage).
5. Patients must be deemed healthy except for diagnosis of ROSAH syndrome and its clinical manifestation.
6. Patients must be at least 18 years of age but no older than 65 years of age at the time of Screening.

Exclusion Criteria:

1. Males who plan to father a child or donate sperm while enrolled in this study or within 90 days after the last dose of study drug.
2. Females who are pregnant, breastfeeding, planning to become pregnant, or planning to donate eggs while on study medication or within 90 days after the last dose of study drug.
3. Use of any of the following prohibited medications:

   * Agents that are known to have systemic anti-inflammatory responses or high risk for nephrotoxicity or hepatotoxicity
   * Moderate CYP3A4 inhibitors: e.g., amiodarone, amprenavir, conivaptan, delavirdine, diltiazem, erythromycin, fluconazole, fosamprenavir, imatinib, miconazole, verapamil, grapefruit juice, cat's claw (Dolichandra unguis-cati), Echinacea augustifolia, wild cherry, chamomile, licorice
   * Strong CYP3A4 inhibitors: e.g., ceritinib, clarithromycin, cobicistat, elvitegravir/ritonavir, idelalisib, indinavir/ritonavir, itraconazole, ketoconazole, lopinavir/ritonavir, nefazodone, nelfinavir, paritaprevir/ritonavir, ombitasvir/paritaprevir/ritonavir (and/or dasabuvir), posaconazole, ritonavir, saquinavir/ritonavir, telithromycin, tipranavir/ritonavir, voriconazole.
   * Strong CYP3A4 inducers: apalutamide, carbamazepine, enzalutamide, ivosidenib, lumacaftor/ivacaftor, mitotane, phenytoin, rifampin, St. John's wort.
   * Digoxin
   * Agents known to cause Torsade de Pointes: Disopyramide, procainamide, quinidine, sotalol, azithromycin, clarithromycin, erythromycin, ciprofloxacin, levofloxacin, moxifloxacin, fluconazole, ketoconazole, pentamidine, voriconazole, haloperidol, thioridazine, ziprasidone, citalopram, escitalopram, dolasetron, droperidol, granisetron, and ondansetron
   * Investigational agents (small molecules and oligonucleotides), vaccines, or invasive medical devices within 28 days (4 weeks, or 5 half-lives, whichever is longer) prior to enrollment or having received a biological product within 6 months prior to enrollment.
4. History of significant hypersensitivity to products related to DF-003 (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs.
5. Recent (within 3 months prior to screening) or acute changes in the following laboratory values:

   * Platelet count ≤ 120,000/mm3, or
   * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > ULN
   * Bilirubin (total, direct) > ULN or
   * International Normalization Ratio (INR) > ULN, or
   * Serum albumin less than the lower limit of normal, or
   * Estimated creatinine clearance < 70 mL/min/1.73 m2 at Screening, calculated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula, or
   * Hemoglobin A1c (HbA1c) > 8%.
6. Moderate or severe hepatic impairment (categorized as Child-Pugh class B and C, respectively, on the Child-Pugh Score for Cirrhosis Mortality)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Frequency and Severity of Treatment-Emergent Adverse Events (TEAEs) as Assessed by CTCAE v5.0 | Baseline to Day 78 (±2)
Frequency and Severity of Serious Adverse Events (SAEs) (Local and Systemic) as Assessed by CTCAE v5.0 | Baseline to Day 78 (±2)

SECONDARY OUTCOMES:
Eye Uveitis as Measured by Changes in Macular Edema | Baseline, Day 1, Day 2, Day 8 (±2), Day 15 (±2), Day 22 (±2), Day 28 (±2), Day 50 (±2), Day 78 (±2)
Eye Uveitis as Measured by Changes in Optic Nerve Edema | Baseline, Day 1, Day 2, Day 8 (±2), Day 15 (±2), Day 22 (±2), Day 28 (±2), Day 50 (±2), Day 78 (±2)
Eye Uveitis as Measured by Changes in Retinal Vasculitis | Baseline, Day 1, Day 2, Day 8 (±2), Day 15 (±2), Day 22 (±2), Day 28 (±2), Day 50 (±2), Day 78 (±2)
Eye Uveitis as Measured by Changes in Retinal Vascular Leakage | Baseline, Day 1, Day 2, Day 8 (±2), Day 15 (±2), Day 22 (±2), Day 28 (±2), Day 50 (±2), Day 78 (±2)
Changes in Serum Chemokine Levels | Day 1 (±30 minutes prior to dosing), Day 29 (24 hours relative to dosing on Day 28), and Day 78 (approximately same time as Day 29 collection)
  Chemokine (C-C motif) ligand CCL2, CCL4, C-X-C motif chemokine ligand (CXCL)-1, CXCL9, CXCL10
Changes in Serum Cytokine Levels | Day 1 (±30 minutes prior to dosing), Day 29 (24 hours relative to dosing on Day 28), and Day 78 (approximately same time as Day 29 collection)
  Interleukin (IL)-1b, IL-6, IL-8, IL-10, IL-2RA soluble, IL-18, Tumor Necrosis Factor (TNF)-Alpha
Changes in Serum Serum Amyloid A (SAA) Levels | Day 1 (±30 minutes prior to dosing), Day 29 (24 hours relative to dosing on Day 28), and Day 78 (approximately same time as Day 29 collection)
  Serum Amyloid A (SAA) proteins are a family of apolipoproteins associated with high-density lipoprotein (HDL) in plasma
Changes in Serum High-Sensitivity C-reactive Protein (hs-CRP) Levels | Day 1 (±30 minutes prior to dosing), Day 29 (24 hours relative to dosing on Day 28), and Day 78 (approximately same time as Day 29 collection)
Maximum Plasma Concentration (Cmax) of DF-003 | Day 1 (-1, 0.5, 1, 2, 4, 6, 8, and 12 hours relative to dosing), 2 (24 hours post-dose), 8(±2), 15(±2), 22(±2), 28(±2; -1, 0.5, 1, 2, 4, 6, 8, and 12 hours relative to dosing), 29(±2; 24 hours post-dose), 36(±2), 50(±2), 64(±2), 78(±2)
Time to Reach Maximum Plasma Concentration (Tmax) of DF-003 | Day 1 (-1, 0.5, 1, 2, 4, 6, 8, and 12 hours relative to dosing), 2 (24 hours post-dose), 8(±2), 15(±2), 22(±2), 28(±2; -1, 0.5, 1, 2, 4, 6, 8, and 12 hours relative to dosing), 29(±2; 24 hours post-dose), 36(±2), 50(±2), 64(±2), 78(±2)
Area Under the Concentration-Time Curve (AUC) of DF-003 from time zero to time t (AUC0-t) | Day 1 (-1, 0.5, 1, 2, 4, 6, 8, and 12 hours relative to dosing), 2 (24 hours post-dose), 8(±2), 15(±2), 22(±2), 28(±2; -1, 0.5, 1, 2, 4, 6, 8, and 12 hours relative to dosing), 29(±2; 24 hours post-dose), 36(±2), 50(±2), 64(±2), 78(±2)
Area Under the Concentration-Time Curve (AUC) of DF-003 from time zero to the time of the last quantifiable concentration (AUC0-last) | Day 1 (-1, 0.5, 1, 2, 4, 6, 8, and 12 hours relative to dosing), 2 (24 hours post-dose), 8(±2), 15(±2), 22(±2), 28(±2; -1, 0.5, 1, 2, 4, 6, 8, and 12 hours relative to dosing), 29(±2; 24 hours post-dose), 36(±2), 50(±2), 64(±2), 78(±2)
Area Under the Concentration-Time Curve (AUC) of DF-003 from time zero to infinity (AUC0-inf, first dose only) | Day 1 (-1, 0.5, 1, 2, 4, 6, 8, and 12 hours relative to dosing), 2 (24 hours post-dose), 8(±2), 15(±2), 22(±2), 28(±2; -1, 0.5, 1, 2, 4, 6, 8, and 12 hours relative to dosing), 29(±2; 24 hours post-dose), 36(±2), 50(±2), 64(±2), 78(±2)
Terminal Phase Half-Life (t1/2) | Day 1 (-1, 0.5, 1, 2, 4, 6, 8, and 12 hours relative to dosing), 2 (24 hours post-dose), 8(±2), 15(±2), 22(±2), 28(±2; -1, 0.5, 1, 2, 4, 6, 8, and 12 hours relative to dosing), 29(±2; 24 hours post-dose), 36(±2), 50(±2), 64(±2), 78(±2)

OTHER OUTCOMES:
Changes in Eye Anterior Chamber Aqueous Fluid Chemokine Levels | Day 1 (±30 minutes prior to dosing), Day 29 (24 hours relative to dosing on Day 28), and Day 78 (approximately same time as Day 29 collection)
  Eye anterior chamber fluid collection is optional and will be collected for assessment of chemokine (C-C motif) ligand CCL2, CCL3, CCL4, CCL5, C-X-C motif chemokine ligand (CXCL)-1, CXCL9, CXCL10
Changes in Eye Anterior Chamber Aqueous Fluid Cytokine Levels | Day 1 (±30 minutes prior to dosing), Day 29 (24 hours relative to dosing on Day 28), and Day 78 (approximately same time as Day 29 collection)
  Eye anterior chamber fluid collection is optional and will be collected for assessment of Interleukin (IL)-1b, IL-6, IL-8, IL-10, IL-2RA soluble, IL-18, Tumor Necrosis Factor (TNF)-Alpha, Serum Amyloid A (SAA), and high-sensitivity C-reactive protein (hs-CRP) levels
Changes in Eye Anterior Chamber Aqueous Fluid Serum Amyloid A (SAA) Levels | Day 1 (±30 minutes prior to dosing), Day 29 (24 hours relative to dosing on Day 28), and Day 78 (approximately same time as Day 29 collection)
  Eye anterior chamber fluid collection is optional and will be collected for assessment of Serum Amyloid A (SAA), and high-sensitivity C-reactive protein (hs-CRP) levels
Changes in Eye Anterior Chamber Aqueous Fluid High-Sensitivity C-reactive protein (hs-CRP) levels | Day 1 (±30 minutes prior to dosing), Day 29 (24 hours relative to dosing on Day 28), and Day 78 (approximately same time as Day 29 collection)
  Eye anterior chamber fluid collection is optional and will be collected for assessment of high-sensitivity C-reactive protein (hs-CRP) levels
Change in Headache Impact Test-6 (HIT-6) Scores | Baseline to Day 28 (±2)
  To evaluate the effects of DF-003 on headache in ROSAH syndrome patients. Test scores range from 36 to 78, with larger scores reflecting greater impact. Little or no impact = HIT-6 score of 49 or less; some impact = HIT-6 score of 50-55; substantial impact = HIT-6 score of 56-59; severe impact = HIT-6 score > 60.
Change in EuroQol 5 Dimension 5 Level (EQ-5D-5L) Scores | Baseline to Day 28 (±2)
  To evaluate the effects of DF-003 on health-related quality of life in ROSAH syndrome patients. This test assesses frequency of symptoms on a 7-point scale (0=no impairment, 6=maximum impairment).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Duke Eye Center - Duke University Hospital, Durham, North Carolina
  - John A. Moran Eye Center - University of Utah Health, Salt Lake City, Utah
- Save Sight Institute - University of Sydney Eye Hospital, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No